CLINICAL TRIAL: NCT06733025
Title: The Effectiveness of Spasticity-correcting Upper Limb Surgery Versus Botulinum Toxin Injections in Patients With Upper Limb Spasticity: an Experimental Study With Paired Design
Brief Title: Comparing Upper Limb Surgery and Botulinum Toxin for Spasticity: A Paired Design Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Promobilia Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Etik_Dnr 2024-05157-01
Record Dates: First submitted 2024-12-09; First posted 2024-12-13 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2024-12

CONDITIONS: Muscle Spasticity; Spinal Cord Injury; Stroke; Traumatic Brain Injuries
Keywords: Muscle spasticity; spinal cord injury; stroke; traumatic brain injuries; tendon lengthening; Botulinum toxin injection
MeSH Terms: conditions — Muscle Spasticity; Spinal Cord Injuries; Stroke; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BoNT injection (Experimental): The participants will first receive BoNT injection for their upper limb spasticity. Earliest three months after the injection they will undergo surgery.
  Interventions: Drug: BoNT Injections
- Surgery (Experimental)
  Interventions: Procedure: Tendon lengthening surgery

INTERVENTIONS:
Procedure: Tendon lengthening surgery — The participants will first receive BoNT injections, earliest three months after they will undergo tendon lengthening surgery
  Arms: Surgery
Drug: BoNT Injections — The dosage and number of injected muscles will vary depending on the degree and extent of spasticity. All patients had previous BoNT injections, one injection circle will be followed in this study.
  Arms: BoNT injection

SUMMARY:
Spasticity is a common complication following central nervous system injuries. Left untreated, spasticity can lead to various complications, hindering activities of daily living and diminishing independence. Spasticity affecting the hand is particularly debilitating because it prevents prehension and grasp, which are critical factors for the ability to perform activities of daily living independently. Spasticity is described as one of the prominent secondary conditions in individuals with various disabilities.

While Botulinum toxin(BoNT) injections are widely used for focal spasticity, surgical interventions remain underutilized despite promising long-term outcomes. Center for Advanced Reconstruction of Extremities(C.A.R.E), at the hand surgery department at Sahlgrenska University hospital in Gothenburg, Sweden is a multiprofessional team and advocates a stratified surgical algorithm based on residual motor function, aiming to optimize patient outcomes.

This open-label, non-randomized, paired study aims to compare the efficacy of spasticity-correcting upper limb surgery with BoNT injections in improving body function, activity, and participation in patients with upper limb spasticity. A total of 30 patients will undergo both interventions sequentially, allowing for within-patient comparisons. The sample size calculation is based on prior studies.

All patients with ongoing BoNT treatment who get referral to C.A.R.E and seem eligible for the study will be informed about the study and enrolment procedure. Eligible participants will undergo both treatments sequentially, with outcome assessments conducted before and after each intervention. The treatments will follow routine clinical care.

The primary outcome measure, Modified Ashworth Scale, will assess spasticity severity. Secondary outcomes will include measures of functional and activity changes specific to each treatment regimen.

This study aims to provide valuable insights into the comparative effectiveness of spasticity interventions, guiding treatment decisions for patients with upper limb spasticity.

DETAILED DESCRIPTION:
Introduction Spasticity is a common secondary complication after injuries to the central nervous system (CNS), and reported in 30% of patients with stroke, 60% of patients with traumatic brain injury (TBI), and 80% of patients with spinal cord injuries (SCI). Spasticity can negatively affect the ability to perform activities. Spasticity affecting the hand is particularly debilitating because it prevents prehension and grasp, which are critical factors for the ability to perform activities of daily living (ADLs) independently. Spasticity is described as one of the prominent secondary conditions in individuals with various disabilities. Previous reviews and studies highlight that future research should focus on improving spasticity management. There is a variation of available treatment options for management of spasticity. Hence, there is conflicting evidence regarding the effectiveness of available spasticity treatments. In many countries, Botulinum toxin (BoNT) injection is considered the gold-standard treatment for focal spasticity. Weak study design and lack of comparative studies between surgery and BoNT holds as reasons why BoNT has displaced surgery. In a recent review of management options for focal spasticity, surgery in the adult population was only recommended in four of thirteen papers. The underutilization of upper limb (UL) surgery has been questioned by surgeons who consider it to be a missed opportunity, especially considering the promising long-lasting results. There is a lack of studies evaluating the effectiveness of alternative treatment approaches for adult patients with UL spasticity after CNS injuries in comparison to the BoNT injections.

Background and rationale Spasticity is a heterogeneous neurological disorder. Treatment goals therefore varies greatly and makes regimen-specific rehabilitation beneficial. The surgical algorithm used at Centre of Advanced Reconstruction of Extremities (C.A.R.E), at Sahlgrenska University hospital (SU) stratifies patients into three different regimens depending on their degree of residual motor function (non-, low-, or high-functioning regimen NFR, LFR, HFR). The rationale for this is that the choice of intervention should be based on whether beneficial gains could be expected after surgery. The algorithm has been presented in detail previously. When comparing outcomes from different treatments the heterogeneity of the population must be considered. The difference between the groups can be caused by selection bias or differences in unobservable characteristics between groups. To investigate whether the outcome differ depending on patient characteristics and assess which of the two treatments; BoNT injection and spasticity-correcting surgery is the most effective in the long term, this study with a paired study design was designed.

Study design and objectives This open-label, non-randomized, experimental paired study aims to investigate the effectiveness of spasticity-correcting UL surgery vs BoNT injections with respect on body function, activity and participation in patients with UL spasticity.

Methods Sample size calculations are based on parameters that have been previously obtained for the primary outcome measure, i.e Modified Ashworth Scale (MAS). MAS showed an average improvement of 1.3 units (SD: 0.7) for surgery, and 0.6 units (SD: 0.5) for treatment with BoNT (11, 14). Assuming a significance level of 0.05, 80% power, SD = 0.7, and an average correlation between repeated measures within patients of 0.5 yields a sample size of 10 patients, or 30 patients as the analyses will be done independently in each of the three regimens.

Study design and participants All patients with ongoing BoNT treatment who get referral to C.A.R.E the hand surgery unit at SU and seem eligible for the study will be informed about the study and enrolment procedure. All individuals who express interest in partaking, will undergo a screening procedure by the Primary Investigator of the study to assess whether they meet the study's eligibility criteria. Study participants will first receive treatment A: BoNT injections in spastic UL muscles. The dosage and number of injected muscles depend on the degree and extent of spasticity and decided by the treating team. To rule out carryover effects earliest three months after the BoNT injections participants receive treatment B. To further rule out the existence of carryover effects from treatment A, new baseline evaluation before treatment B will take place.

Treatment B: spasticity-correcting UL surgery. The degree of tendon lengthening, and number of lengthened muscles depend on the degree and extent of spasticity and decided by the treating team. The patients will be assessed with the same measurement pre-, 4-6 weeks and 3 months after BoNT, as well as before surgery and 6 months after surgery. Eligibility criteria: 1. 18 years or above; 2. Problematic spasticity characterized by a velocity-dependent increase in tonic stretch reflexes or intermittent or sustained involuntary muscle activity in the UL after stroke, TBI or SCI; 3. At least 6 months since the injury event; 4. Ongoing BoNT treatment in the UL; 5. A minimum of 3 months must have passed since the last BoNT injection; 6. At least two muscles in the hand/wrist must be considered suitable for surgical intervention; 7. Medically stable to undergo surgery; 8. No other severe UL injury's that affect the individual's functional level. The study has ethical approval Dnr:2024-05157-01. The study will be conducted in accordance with relevant ethical guidelines.

The primary outcome measure in the whole study population is spasticity measured with Modified Ashworth Scale (MAS). The single-item MAS is measured on a six-point scale from 0 (no increase in muscle tone) to 4 (affected part rigid in flexion or extension), with an additional point allocated at 1+ (slight increase in muscle tone). For analysis purposes, the MAS scores in the treated muscles will be summed to provide a "composite spasticity score".

Treatment A: BoNT injections The BoNT treatment is part of routine care at the tonus clinics at rehabilitation medicine at SU, NU hospital group and Södra Älvsborg hospital (SÄS). All units are specialized in the care of patients with neurological injuries, mainly stroke, SCI and TBI. When injected in spastic muscles, BoNT blocks certain chemical signals from nerves, which results in temporary relaxation of muscles. Normally, the effect wear off after 3 months, and its maximum (peak) effect typically occurs after 4-6 weeks following injection. In the present study, the dosage and number of injected muscles will vary depending on the degree and extent of spasticity. All patients had previous BoNT injections, one injection circle will be followed in this study. Training is allowed directly after the injections. The injections will be given by specialized doctors, with many years of experience of BoNT injections in the study population. Following the BoNT injections, participants will receive standard rehabilitation. This will vary but commonly involve stretching, strength training of the antagonists, and in some cases splinting.

Treatment B: Surgical treatment The surgical treatment is part of routine care at C.A.R.E. the hand surgery unit SU. The spasticity-correcting procedures are performed by a stair-step incision technique followed by reattachment in the lengthened position using a side-to-side, cross-stich technique. The degree of tendon lengthening is decided by aiming for normal resting length, which are estimated at full relaxation during general anesthesia; 2-3 cm are usually sufficient. The day after surgery, wrapping and custom-made splints are fashioned, with the aim to facilitate prolonged soft tissue stretch and prevent postoperative edema. When possible, dynamic activation of the antagonist muscles of the lengthened muscles are performed the first day after surgery, as well as passive or dynamic activation of treated muscles. Active range of motion (ROM) exercises are allowed to the maximum ROM with no restrictions in lengthened muscles, or their antagonists. The rehabilitation protocol has previously been described in detail.

Statistical analysis plan Demographics and baseline characteristics will be summarized using descriptive statistics. Visual inspection of histograms and QQ-plots will be used to graphically check for approximate normality. Descriptive analyses include the graphical presentation of individual trajectories of the primary outcome measure (MAS) over time as well as box plots for the time-dependent distribution of MAS. The individual change in outcome measure after each treatment will be calculated. Mean or median values will be compared by treatment accounting for the paired design of the study, i.e. paired t-test or Wilcoxon signed-rank test for interval or ordinal data, and Mc Nemar's test for binary data. Furthermore, we will use multiple regression to determine which background factors are associated with the two treatment effects separately, and with the difference between treatment effects. Example for background factors: age, sex and regimens.

Clinical relevance The severity of spasticity can vary greatly depending on whether the spasticity is uni- or bilateral and the existence and severity of concomitant CNS syndromes may further add to the severity. The main goal of any spasticity intervention is to improve function, although the treatment potential greatly depends on the motor recovery stage of the UL. Hence, the treatment goals vary from restoring active function to improving passive function and facilitate care of the UL. Spasticity-correcting surgery is shown to produce long-term beneficial results. Today, knowledge is lacking regarding which of the two treatments BoNT injections and spasticity-correcting surgery is most effective in the long-term. Increased knowledge about advantages and disadvantages of these two treatment methods could help in the discussion of realistic expectations and occupational goal setting. Today healthcare lacks the knowledge to convey to patients, decision makers and relatives about the advantages and disadvantages of these two treatment methods, which is why research into the effectiveness of the methods is in demand. If the outcome of comparisons shows that the effect is equivalent, future patients will be able to choose the treatment that seems least demanding to the individual. If the outcome instead shows that one method is more beneficial, it will likely be offered to a greater extent in the future. If the outcome is that different functional gains are achieved with the different methods, the patient's prioritized goals are likely to be decisive for the choice of treatment. Increased knowledge will under all circumstances contribute to the selection of the best individual treatment, following a dialogue between patient and the clinicians. Ultimately, it has the potential to raise awareness of the treatment concepts, as a means to efficiently manage and treat UL spasticity. This may in turn increase the number of referrals and thereby increase the number of patients who achieve long-lasting functional and activity-based gains despite a chronic disorder. The aim in the long term is to ensure that all patients with spasticity problems are offered assessment and information about opportunities to enhance hand function.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or above
2. Problematic spasticity, characterised by a velocity-dependent increase in tonic stretch reflexes or intermittent or sustained involuntary muscle activity in the UL after stroke, TBI, or SCI
3. Patients treated at least 6 months after the injury event
4. Ongoing BoNT treatment in the UL
5. A minimum of 3 months passed since the last BoNT injection
6. At least two muscles in the hand and wrist were considered for treatment
7. For the BoNT group, a community occupational or physical therapist was assigned for post BoNT treatment
8. For the surgery group, medically stable to undergo surgery
9. No other severe UL injuries affecting the functional level

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2029-01-29 (Estimated); Study Completion 2029-06-29 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS). | Baseline BoNT, 5weeks, 3months. Baseline surgery, 6 months
  The single-item Modified Ashworth Scale is a six-point scale from 0 (no increase in muscle tone) to 4 (affected part rigid in flexion or extension), with an additional point allocated at 1+ (slight increase in muscle tone). As such, the Modified Ashworth Scale provides a single score to represent spasticity in a specific movement. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Visual Analogue Scale | Baseline BoNT, 5weeks, 3months. Baseline surgery, 6 months
  Self-rated pain intensity will be measured with a Visual Analogue Scale, the scale goes from 0= no pain, to 10= severe pain. Higher scores mean a worse outcome.
Visual Analogue Scale | Baseline BoNT, 5weeks, 3months. Baseline surgery, 6 months
  Self-rated experienced upper limb spasticity will be measured with a Visual Analogue Scale, the scale goes from 0= no spasticity, to 10= severe spasticity. Higher scores mean a worse outcome.
Active Range Of Motion | Baseline BoNT, 5weeks, 3months. Baseline surgery, 6 months
  In target movements with a hand held goniometer, the goniometer measure the joints range of motion, from 0 to 180 degrees range of motion. Higher scores mean a better outcome.
Passive Range Of Motion | Baseline BoNT, 5weeks, 3months. Baseline surgery, 6 months
  With a hand held goniometer the goniometer measure the joints range of motion, from 0 to 180 degrees range of motion. Higher scores mean a better outcome.
The opening ability of the hand | Baseline BoNT, 5weeks, 3months. Baseline surgery, 6 months
  The capacity to achieve passive and active hand opening will be rated using the following scale: hand closed, ¼ open, ½ open, ¾ open, or fully open. The same grading system will be applied to describe the resting position of the hands. Higher scores mean a better outcome.
Jamar | Baseline BoNT, 5weeks, 3months. Baseline surgery, 6 months
  Maximum handgrip strength will be measured with a hydraulic hand dynamometer (JAMAR® 5030J1, Sammons Preston Rolyan, USA). The dynamometer measure the isometric grip force from 0-90 kg. Higher scores mean a better outcome.
Pinch strength | Baseline BoNT, 5weeks, 3months. Baseline surgery, 6 months
  Maximum pinch grip strength will be measured using a Preston Pinch Gauge (European Bissel Healthcare Ltd., Winchester, England). The scale goes from 0-5kg. Higher scores mean a better outcome.
Grasp and Release Test (GRT) | Baseline BoNT, 5weeks, 3months. Baseline surgery, 6 months
  The ability to grasp, move, and release objects will be measured using the Grasp and Release Test. Assesses the ability to pick up, move, and release six objects of varying sizes, weights and textures using a palmar or lateral grasp. The score is the number of times the participants is able to move each object in 30 seconds. Higher scores mean a better outcome.
The Cylinder Test | Baseline BoNT, 5weeks, 3months. Baseline surgery, 6 months
  The ability to actively and/or passively open one's hand and actively grasp and release a cylindrical object will be measured using a Cylinder Test. The test is divided into five subtests; 1) active cylinder grip-normal, 2) active cylinder grip-adapted, 3) active cylinder grip self-assisted, 4) passive cylinder grip-self-assisted, and 5) passive cylinder grip-examiner-assisted. For each of the subtests we will record the size of the largest cylinder that the participant manages to grasp, lift, and release (Subtests 1-3) or simply hold (Subtests 4 and 5). The cylinder ranges go from 20-150cm. Higher scores mean a better outcome.
Visual Analogue Scale | Baseline BoNT, 5weeks, 3months. Baseline surgery, 6 months
  Self-rated arm and hand function (usefulness) will be measured using the Visual Analogue Scale, the scale goes from 0= no hand function to 10= good hand function. Higher scores mean a better outcome.
Arm-Activity Measure Swedish version | Baseline BoNT, 5weeks, 3months. Baseline surgery, 6 months
  The Arm-Activity Measure questionnaire will be used to capture difficulties in passive and active real-life arm functions. The questionnaire asks about the perceived amount of difficulty experiencing doing different tasks, the scale gos from 0= no difficulty to 4= unable to do. The Arm-Activity Measure subscale A range from 0-32 points, The Arm-Activity Measure subscale B goes from 0-52p. Higher scores mean a worse outcome.
Canadian Occupational Performance Measure (COPM) | Baseline BoNT, 5weeks, 3months. Baseline surgery, 6 months
  Limitations in the prioritized daily activities will be measured using the Canadian Occupational Performance Measure. The participant is asked to identify a number of activities of difficulty. They pick out the 5 most important. Theese five activities are scored. The Canadian Occupational Performance Measure, has two main scoring categories which include performance and satisfaction, both are out of 10 points (1-10). A lower score indicates low performance and satisfaction, and a higher score indicates higher performance and satisfaction levels. Higher scores mean a better outcome.
EuroQol five-dimension questionnaire (EQ5D 5 L) | Baseline BoNT, 5weeks, 3months. Baseline surgery, 6 months
  The patients' health-related quality of lifec will be assessed using the EuroQol five-dimension questionnaire.
  The questionnaire include five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. The digits for the five dimensions can be combined into a number that describes the patient's health state. Higher scores mean a worse outcome.
  The EuroQol visual analogue scale records the patient's self-rated health on a vertical visual analogue scale where the endpoints (0-100) are labelled 'The best health you can imagine'(100) and 'The worst health you can imagine'(0). Higher scores mean a better outcome.
Visual Analogue Scale | Baseline BoNT, 5weeks, 3months. Baseline surgery, 6 months
  Self-rated arm and hand cosmetics will be measured using a Visual Analogue Scale, the scale goes from 0= no problem with the look of the upper limb, to 10= severe problem with the look of the upper limb. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hoispital, Mölndal, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
The IDP contains personal goals, performance evaluations, and development needs that are confidential. Sharing it might breach privacy.